CLINICAL TRIAL: NCT05130749
Title: Infection Prevention and Control Practices Among Primary Healthcare Nurses Regarding COVID-19 in Saudi Arabia
Brief Title: Infection Prevention and Control Practices Regarding COVID-19
Acronym: IPCP
Status: Completed | Type: Observational
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Ayat Zammar, Principal Investigator, King Saud University
Other Study IDs: KSU-HE-21-35
Record Dates: First submitted 2021-11-16; First posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: COVID-19 Pandemic
Keywords: Infection Prevention; Infection control; Primary Healthcare; Nurses; Saudi Arabia
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary Healthcare Nurses: Nurses allocated in primary Healthcare settings
  Interventions: Other: Questionnaire
- Non Nurses Primary Healthcare: Other Healthcare providers allocated in primary health care settings
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — The questionnaire's first section asked for demographic information such as gender, age, the name of the primary healthcare centre, and level of education. The second section comprised sources of knowledge on COVID-19; respondents replied on a scale of 1 least used (1), occasionally (2), more frequently (3), and most used (4). The third section had six items pertaining to nurses' infection prevention and control methods with reference to COVID-19, and respondents replied on a scale of yes (2), occasionally (1), and no (0). Permission to use the questionnaire has been requested from the author and is awaited.

SUMMARY:
Background: Healthcare providers, particularly nurses, are at risk of infection as part of the COVID-19 epidemic chain since they assist in the disease's containment. By recognising the risk factors for infection and implementing suitable measures to reduce these risks, all reasonable efforts should be taken to control the spread of infection to them. The major aim of the present study was to determine the level of infection prevention and control practises used by primary healthcare nurses in Saudi Arabia during the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Male and female healthcare practitioners with at least one year of experience and who worked in all areas of primary healthcare facilities during the COVID-19 epidemic.

Exclusion Criteria:

* Healthcare providers that are unwilling to participate in the present study have been eliminated

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: healthcare practitioners and community health nurses who worked at the aforementioned centres. There are 800 nurses in total.
Sampling Method: Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Distribution of study participants by gender, age group, marital status, and income level in a self-reported questionnaire. | Once within 6 weeks
  Demographic data included age, gender, experience, educational level, marital status, income and job will be assessed using numerical code for each demographic variable.

SECONDARY OUTCOMES:
Detection of source of knowledge regarding COVID-19 prevention methods | Once within 6 weeks
  Using self-reporting questionnaire, will assess Social Media, Radio & television, Seminars & workshops, Posters & Pamphlets, Newspapers &Magazines and Seniors & Other Colleagues from (Least used= 1 to Most used= 4).

OTHER OUTCOMES:
Circumstances when Healthcare providers practice infection prevention tasks in settings. | Once within 6 weeks
  Assess the use of Personl Protective Equipments (Gloves, Mask(regular), N95 respirator mask, Surgical mask, Goggles, Apron, Gown, Isolation gown, Hair cover, Shoe cover and Eye protection) from Never(0) to Always (4).

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT05130749/Prot_SAP_000.pdf